CLINICAL TRIAL: NCT00432627
Title: An Open-label, Single-dose, Parallel-group Study to Assess the Pharmacokinetics of 20 mg/kg Oral Deferasirox in Patients With Impaired Hepatic Function and Healthy Subjects With Normal Hepatic Function
Brief Title: Impact of Hepatic Impairment on the Pharmacokinetics of Deferasirox.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2125
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; adults; deferasirox
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild hepatic impaired (Experimental)
  Interventions: Drug: Deferasirox
- Moderate hepatic impaired (Experimental)
  Interventions: Drug: Deferasirox
- Severe hepatic impaired (Experimental)
  Interventions: Drug: Deferasirox
- Healthy volunteers (Experimental): Controlled group
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — one dose of 20 mg/kg/day
  Other Names: ICL670

SUMMARY:
This study is to assess the pharmacokinetics of deferasirox in hepatically impaired patients compared to healthy volunteers.

ELIGIBILITY:
Inclusion criteria for those with hepatic impairment:

* Physical signs consistent with a clinical diagnosis of liver cirrhosis
* Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment
* Otherwise considered healthy

Inclusion criteria for healthy volunteers:

• In good health.

Exclusion criteria for those with hepatic impairment:

* Clinically significant abnormal findings other than hepatic impairment
* Clinical evidence of severe ascites
* History of surgical portosystemic shunt
* Any evidence of progressive liver disease within the last 4 weeks

Exclusion criteria for healthy controls:

* Clinical evidence of liver disease or liver injury
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result
* Use of any prescription medication within 1 month prior to dosing

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of deferasirox and its metabolites | at FPFV and at LPLV

SECONDARY OUTCOMES:
Safety and tolerability of deferasirox assessed by adverse events | at FPFV and at LPLV

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Kiel, Germany

REFERENCES:
- See also: Results can be found for CICL670A2125 on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4382